CLINICAL TRIAL: NCT01585662
Title: Random Comparing Study on Two Different EUS-guided Pseudocyst Drainage Methods--Modified Naso-pancreatic Tube Drainage and Stents Drainage
Brief Title: Prospective Random Comparing Study on EUS-guided Pseudocyst Drainage by Naso-pancreatic Tube and Stents
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoyin Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaoyin Zhang, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2012-04-19; First posted 2012-04-26 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Pseudocyst
Keywords: EUS; pancreatic pseudocyst; drainage
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naso-pancreatic tube (Experimental): The patients enrolled in this group will be treated with modified naso-pancreatic tube drainage method.
  Interventions: Procedure: EUS-guided pancreatic pseudocyst drainage
- Stents (Experimental): The patients enrolled this group will be treated by placing the stents (at least 2 stents) between gastric and pancreatic pseudocyst.
  Interventions: Procedure: EUS-guided pancreatic pseudocyst drainage

INTERVENTIONS:
Procedure: EUS-guided pancreatic pseudocyst drainage — EUS-guided pancreatic pseudocyst drainage by one 8 French naso-pancreatic tube or 2-3 two pig tails- stents.
  Other Names: Naso-pancreatic drainage tube:8 Fren,made by Cook Company; Two pig tails- stents:5cm long,made by Cook Company

SUMMARY:
EUS-guided pseudocyst drainage has been used world widely. Now, most endoscopists tend to place several stents to drain the content of cyst into GI tract. In the investigators experience, a modified naso-pancreatic tube drainage was more safer, easier and cheaper than placement of stents. Moreover, none of pseudocysts(total 19) drained by this modified naso-pancreatic tube drainage method were found recurrent with a follow up period from 3 months-34 months. So, the investigators designed this prospective random comparing study to confirm the result.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with ages from 18-80 years old.
2. The pseudocysts were formed more than 3 months.
3. The size of pseudocyst is more than 5 cm.
4. The patient has the symptoms related with the pseudocyst.
5. The distance between gastric and the wall of the pseudocyst is less than 1 cm from CT image.
6. The consent form has been signed.

Exclusion Criteria:

1. The patient can't accept the endoscopic procedure.
2. The patient has blood coagulation dysfunction.
3. The patient has mental disorders.
4. The patient has mild or severe cardiorespiratory insufficiency.
5. The patient has hypertension and can't be controlled to safe level.
6. Diabetics whose blood sugar level can't be controlled to safe level.
7. Patients with alcohol dependence
8. Pregnant and lactating women.
9. The patients the investigator don't think suitable for this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of pancreatic pseudocyst | 12 months

SECONDARY OUTCOMES:
The complication rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wu Kaichun, MD,PhD, Study Chair — The forth military medical university
Locations (1):
- Xijing Institute of digestive diseases, Xian City, Shanxi, China

REFERENCES:
- [Background] Baron TH, Wiersema MJ. EUS-guided transesophageal pancreatic pseudocyst drainage. Gastrointest Endosc. 2000 Oct;52(4):545-9. doi: 10.1067/mge.2000.108928. No abstract available. PMID 11023579
- [Background] Seewald S, Thonke F, Ang TL, Omar S, Seitz U, Groth S, Zhong Y, Yekebas E, Izbicki J, Soehendra N. One-step, simultaneous double-wire technique facilitates pancreatic pseudocyst and abscess drainage (with videos). Gastrointest Endosc. 2006 Nov;64(5):805-8. doi: 10.1016/j.gie.2006.07.049. PMID 17055880
- [Background] Lopes CV, Pesenti C, Bories E, Caillol F, Giovannini M. Endoscopic-ultrasound-guided endoscopic transmural drainage of pancreatic pseudocysts and abscesses. Scand J Gastroenterol. 2007 Apr;42(4):524-9. doi: 10.1080/00365520601065093. PMID 17454865
- [Background] Barthet M, Lamblin G, Gasmi M, Vitton V, Desjeux A, Grimaud JC. Clinical usefulness of a treatment algorithm for pancreatic pseudocysts. Gastrointest Endosc. 2008 Feb;67(2):245-52. doi: 10.1016/j.gie.2007.06.014. PMID 18226686